CLINICAL TRIAL: NCT02171078
Title: Post-Treatment Surveillance in Breast Cancer: Bringing Cost Effectiveness Research (CER) to the Alliance
Brief Title: Post-Treatment Surveillance in Breast Cancer: Bringing CER to the Alliance
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); American College of Surgeons (Other); Alliance for Clinical Trials in Oncology (Other); Harvard University (Other); Dana-Farber Cancer Institute (Other); M.D. Anderson Cancer Center (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0742; CE-1304-6543 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute); UW14041 (Other: University of Wisconsin Carbone Cancer Center); A539713 (Other: UW Madison); SMPH/SURGERY/SURG ONC (Other: UW Madison)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Breast Neoplasms; Health Services Research; Surveillance; Diagnostic Imaging; Magnetic Resonance Imaging; Mammography; Toxicity; Adverse Effects; Side Effects; Recurrence
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alliance for Clinical Trials Database: Use existing data from clinical trials sponsored by one of the leading cancer cooperative groups to evaluate how risk of recurrence and side effects of treatment vary based on patient and cancer characteristics.
- National Cancer Database: Use existing data to evaluate the effectiveness of the latest imaging technology for detecting recurrence and improving survival in patients previously treated for breast cancer.
- Stakeholder Engagement: Engage cancer survivors, providers, and health outcomes researchers in the development of an improved patient-centered approach to guide post-treatment care, as well as identification of the highest priority strategies for prospective randomized trials.

SUMMARY:
Nearly three million living women have survived breast cancer. Physicians rely on clinical practice guidelines to make decisions on follow-up care. Among other things, the goal is to monitor for recurrence or side effects of treatment among survivors. It is unclear whether these guidelines represent the best approach for any given patient as they do not account for differences in disease or patient preferences and may not consider recent advances in imaging and treatment options. We seek to develop a new approach to surveillance following breast cancer treatment which will be more patient-centered and effective than the existing one-size-fits-all approach and will consider individual risk factors.

DETAILED DESCRIPTION:
Our project involves three primary goals:

1. Use existing data from clinical trials sponsored by one of the leading cancer cooperative groups to evaluate how risk of recurrence and side effects of treatment vary based on patient and cancer characteristics.
2. Use existing data to evaluate the effectiveness of the latest imaging technology for improving survival in patients previously treated for breast cancer.
3. Engage cancer survivors, providers, and health outcomes researchers in the development of an improved patient-centered approach to guide post-treatment care, as well as identification of the highest priority strategies for prospective randomized trials.

Methods Our methods have been developed based on input from patients and other stakeholders who identified the need for a large-scale observational study. The goal is to produce timely results, and guide the development of an improved approach to surveillance that recognizes individual patient risk factors and allows for design of future prospective studies. This study analyzes recurrence data and treatment side effects on over 22,000 patients involved in past clinical trials on breast cancer care. The project also involves the analysis of existing data (n=15,000 patients) from a national cancer registry (National Cancer Database) to evaluate whether new imaging technology, beyond mammography, are able to detect recurrence earlier and improve survival. Finally, we will engage cancer survivors, health care providers, and researchers to develop new guidance for the care and monitoring of breast cancer survivors, and to guide and prioritize future prospective trials.

ELIGIBILITY:
Inclusion Criteria:

* Women (all Aims)
* Diagnosis of breast cancer (Aims 1 & 2)
* American Joint Committee on Cancer (AJCC) stages I-III (Aim 1) AJCC stages II-III (Aim 2)
* Patient, health care provider, and researcher stakeholders (Aim 3)

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Research Aim 1: Patients who have participated in 1 of 15 closed clinical trials; Research Aim 2: National Cancer Database (NCDB); Research Aim 3: Purposive sample of breast cancer survivor, breast cancer treatment provider, and cancer health services researcher stakeholders
Sampling Method: Non-Probability Sample
Enrollment: 34359 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Time to Recurrence | 5 Years from Diagnosis
  Data elements include the date and site of recurrence, type of recurrence (e.g., local/regional or distant recurrence), and progression.
Time to Toxicity/Side Effects of Treatment | Within relevant timeframe of legacy clinical trial. Most trials include 2-year follow-up
  Legacy clinical trials contain detailed data on treatment toxicity and complications. Most trials include 2-year follow-up to determine the prevalence and time to presentation for each of the following toxicities: lymphedema, cardiotoxicity, and pneumonitis
  Safety Issue?:
  No

SECONDARY OUTCOMES:
Time to Death | Within 5 years from time of diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Caprice C Greenberg, MD MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Result] Schumacher JR, Neuman HB, Yu M, Vanness DJ, Si Y, Burnside ES, Ruddy KJ, Partridge AH, Schrag D, Edge SB, Zhang Y, Jacobs EA, Havlena J, Francescatti AB, Winchester DP, McKellar DP, Spears PA, Kozower BD, Chang GJ, Greenberg CC; Alliance ACS-CRP CCDR Breast Cancer Surveillance Working Group. Surveillance Imaging vs Symptomatic Recurrence Detection and Survival in Stage II-III Breast Cancer (AFT-01). J Natl Cancer Inst. 2022 Oct 6;114(10):1371-1379. doi: 10.1093/jnci/djac131. PMID 35913454
- [Result] Schumacher JR, Wiener AA, Greenberg CC, Hanlon B, Edge SB, Ruddy KJ, Partridge AH, Le-Rademacher JG, Yu M, Vanness DJ, Yang DY, Havlena J, Strand C, Neuman HB. Local/Regional Recurrence Rates After Breast-Conserving Therapy in Patients Enrolled in Legacy Trials of the Alliance for Clinical Trials in Oncology (AFT-01). Ann Surg. 2023 May 1;277(5):841-845. doi: 10.1097/SLA.0000000000005776. Epub 2022 Dec 14. PMID 36521077
- [Result] Dudley CM, Wiener AA, Stankowski-Drengler TJ, Schumacher JR, Francescatti AB, Poore SO, Greenberg CC, Neuman HB. Rates of Ipsilateral Local-regional Recurrence in High-risk Patients Undergoing Immediate Post-mastectomy Reconstruction (AFT-01). Clin Breast Cancer. 2021 Oct;21(5):433-439. doi: 10.1016/j.clbc.2021.03.009. Epub 2021 Mar 27. PMID 34103255
- [Result] Adesoye T, Schumacher J, Greenberg CC. ASO Author Reflections: Use of Breast Imaging After Treatment for Locoregional Breast Cancer (AFT-01). Ann Surg Oncol. 2019 Dec;26(Suppl 3):553-554. doi: 10.1245/s10434-018-7070-9. Epub 2018 Dec 18. No abstract available. PMID 30565039
- [Result] Wong ML, McMurry TL, Schumacher JR, Hu CY, Stukenborg GJ, Francescatti AB, Greenberg CC, Chang GJ, McKellar DP, Walter LC, Kozower BD. Comorbidity Assessment in the National Cancer Database for Patients With Surgically Resected Breast, Colorectal, or Lung Cancer (AFT-01, -02, -03). J Oncol Pract. 2018 Oct;14(10):e631-e643. doi: 10.1200/JOP.18.00175. Epub 2018 Sep 12. PMID 30207852
- [Derived] Krecko LK, Neuman HB, Greenberg CC, Wilke LG, Hanlon BM, Edge SB, Ruddy KJ, Partridge AH, Le-Rademacher J, Yang DY, Havlena J, R Schumacher J. Validation of the AJCC 8th Edition Breast Cancer Prognostic Staging System in Legacy Alliance Trials (AFT-01). Ann Surg Oncol. 2024 Sep;31(9):5880-5887. doi: 10.1245/s10434-024-15477-5. Epub 2024 Jun 2. PMID 38825628
- [Derived] Neuman HB, Schumacher JR, Edge SB, Ruddy KJ, Partridge AH, Yu M, Vanness DJ, Hanlon BM, Le-Rademacher JG, Yang DY, Havlena J, Strand CA, Greenberg CC. The influence of anatomic stage and receptor status on first recurrence for breast cancer within 5 years (AFT-01). Cancer. 2023 May 1;129(9):1351-1360. doi: 10.1002/cncr.34656. Epub 2023 Mar 6. PMID 36872873
- [Derived] Stankowski-Drengler TJ, Schumacher JR, Hanlon B, Livingston-Rosanoff D, Van de Walle K, Greenberg CC, Wilke LG, Neuman HB. Outcomes for Patients with Residual Stage II/III Breast Cancer Following Neoadjuvant Chemotherapy (AFT-01). Ann Surg Oncol. 2020 Mar;27(3):637-644. doi: 10.1245/s10434-019-07846-2. Epub 2020 Jan 3. PMID 31900808
- [Derived] Schumacher JR, Neuman HB, Chang GJ, Kozower BD, Edge SB, Yu M, Vanness DJ, Si Y, Jacobs EA, Francescatti AB, Spears PA, Havlena J, Adesoye T, McKellar D, Winchester D, Burnside ES, Greenberg CC; Alliance ACS-CRP CCDR Breast Cancer Surveillance Working Group. A National Study of the Use of Asymptomatic Systemic Imaging for Surveillance Following Breast Cancer Treatment (AFT-01). Ann Surg Oncol. 2018 Sep;25(9):2587-2595. doi: 10.1245/s10434-018-6496-4. Epub 2018 May 17. PMID 29777402
- [Derived] Adesoye T, Schumacher JR, Neuman HB, Edge S, McKellar D, Winchester DP, Francescatti AB, Greenberg CC; Alliance ACS-CRP CCDR Breast Cancer Surveillance Working Group. Use of Breast Imaging After Treatment for Locoregional Breast Cancer (AFT-01). Ann Surg Oncol. 2018 Jun;25(6):1502-1511. doi: 10.1245/s10434-018-6359-z. Epub 2018 Feb 15. PMID 29450753
- [Derived] Neuman HB, Schumacher JR, Francescatti AB, Adesoye T, Edge SB, Vanness DJ, Yu M, McKellar D, Winchester DP, Greenberg CC; Alliance/American College of Surgeons Clinical Research Program Cancer Care Delivery Research Breast Cancer Surveillance Working Group. Risk of Synchronous Distant Recurrence at Time of Locoregional Recurrence in Patients With Stage II and III Breast Cancer (AFT-01). J Clin Oncol. 2018 Apr 1;36(10):975-980. doi: 10.1200/JCO.2017.75.5389. Epub 2018 Jan 31. PMID 29384721
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/